CLINICAL TRIAL: NCT02053935
Title: Impact of Dopamine Infusion on Insulin Secretion in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Rubina Heptulla, Division Chief of Pediatric Endocrinology, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-286
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Hyperglycemia; Sepsis
Keywords: Dopamine; hyperglycemic clamp; sepsis; hyperglycemia; insulin secretion
MeSH Terms: conditions — Hyperglycemia; Sepsis | interventions — Dopamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dopamine (Other): All patients will receive the same intervention.
  Interventions: Drug: Dopamine

INTERVENTIONS:
Drug: Dopamine — Each subject will receive a priming dose of dextrose 20% to increase their glucose concentration by 125 mg/dl in the first 15 minutes. Then they will receive variable rates of dextrose 20% infusion to maintain glucose level at 180-220 mg/dl. Then, dopamine (200mg/250ml) will be titrated up to 5 mcg/kg/min with care not to increase blood pressure greater than 160 systolic. Dopamine will be infused for 3 hours.

SUMMARY:
This is a clinical study of a drug named dopamine and how it affects our bodies ability to make and secrete insulin. Insulin is a hormone made in the pancreas that helps our body regulate sugar levels. We think that this drug decreases the amount of insulin our body makes and causes our sugar levels to be high. When you are critically ill there can be many adverse effects if you have sugar levels that are too high.

DETAILED DESCRIPTION:
Rationale Role of dopamine infusion on pancreatic beta cell function in health and disease remain undetermined in humans. Increasingly, hyperglycemia in the critical care arena bodes poorly on health outcomes.

This study for the first time investigates the role of dopamine infusion in health and has the potential to guide larger studies on impact of dopamine use in critical illness.

Study Design This project will be a prospective, single-center trial to determine the effect of dopamine in healthy subjects using the hyperglycemic clamp.

Study Procedures:

After signing informed consent subjects will undergo screening at the clinical research center after an overnight fast. At this visit, a complete history and physical exam including vital signs, height, weight, BMI, waist circumference will be obtained. Cardiac conditions will be screened using an EKG. Baseline labs will be drawn at this visit, including CBC, chemistry, liver function tests, hemoglobin AIC, thyroid function tests, lipids and cortisol. Females will have a urine beta HCG.

Subjects that meet study criteria will return within 30 days of screening to the clinical research after an overnight fast. One large bore (20 gauge) venous cannula will be inserted in the antecubital fossa for infusion of dopamine and dextrose 20% intravenous solution. Another cannula will be inserted in the contralateral arm for frequent blood sampling.

Insulin sensitivity will be determined using the gold standard hyperglycemic clamp as previously described (DeFronzo, 1979).13 Each subject will act as their own control and receive placebo infusion followed by dopamine infusions.

Subjects will have their blood pressure, heart rate, and glucose monitored every 10 minutes. Each subject will receive a priming dose of dextrose 20% to increase their glucose concentration by 125 mg/dl in the first 15 minutes. Then they will receive variable rates of dextrose 20% infusion to maintain glucose level at 180-220 mg/dl. C-peptide, insulin, glucagon and catecholamine levels will be drawn at 30 min and 60 min to determine baseline levels prior to dopamine infusion. Then, dopamine (200mg/250ml) will be titrated up to 5 mcg/kg/min with care not to increase blood pressure greater than 160 systolic. C-peptide, insulin level, glucagon, plasma catecholamines will be measured at 90 min and 120 min, 150min, 180min, 210min, 240min. At 120min, 180 min and 240 min glucagon and cortisol levels will also be measured. The total amount of blood withdrawn for entire study will be less than 100 ml. After all blood samples are drawn, dextrose and dopamine infusion will be down-titrated and stopped. The subject will be given lunch and glucose level will be checked. Venous cannulas will then be removed and subject will be sent home.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects
2. Age 18-35 years
3. Hemoglobin >12 g/dl
4. Euthyroid or on a stable dose of synthroid
5. Normal EKG, hemoglobin AIC, kidney and liver function

Exclusion Criteria:

1. Prior history of dopamine infusion
2. Past medical history of diabetes, hypertension, myocardial infarction, vaso-occlusive disease or arrhythmias
3. Chronic steroid therapy, oral contraceptive pills, monoamine oxidase inhibitors (MAO-I), anticonvulsants (phenytoin)
4. Pregnant women because dopamine is pregnancy category C
5. Clinical signs of polycystic ovarian syndrome
6. Past medical history of Cushing's disease or pheochromocytoma
7. Sulfa drug allergy
8. Use of any medications or illness determined by the investigators that may affect insulin secretion or insulin sensitivity.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
insulin secretion | 4 hours
  Insulin secretion will be assessed via glucose infusion requirement during a hyperglycemic clamp. Insulin and c-peptide levels will be monitored. Insulin secretion will be attenuated by 30% from baseline in subjects receiving dopamine

SECONDARY OUTCOMES:
counter-regulatory hormones | 4 hours
  Counter-regulatory hormone concentrations before, during and after dopamine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Erika Mark, DO, Study Director — Albert Einstein College of Medicine; Rubina Heptulla, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center of Albert Einstein College of Medicine, The Bronx, New York, United States